CLINICAL TRIAL: NCT06861907
Title: IMPRINT Randomized Evaluation
Brief Title: IMPRINT VR Trainer Evaluation
Status: Completed | Type: Observational
Sponsor: Charles River Analytics (Industry)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH); The New England Consortium (Unknown)
Responsible Party: Principal Investigator, E Vincent Cross, Senior Research Scientist, Charles River Analytics
Other Study IDs: CharlesRiverA; 2R44ES031818-02 (NIH)
Record Dates: First submitted 2025-02-26; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Virtual Reality
Keywords: HAZWOPER; HAZMAT; Training; Virtual Reality

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trainers: Trainers responsible to teaching the 40-hr HAZWOPER course. They are experts in their field and have the most familiarity with the traditional PowerPoint training
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Virtual Reality Modules created to simulate HAZWOPER PowerPoint scenarios

SUMMARY:
The goal of this study is to assess whether the Immersive Modular Preparedness Intelligent Tutor (IMPRINT) virtual reality (VR) training modules provide a measurable benefit in training delivery and trainee engagement. Specifically, the investigators want to see how VR can enhance trainees' comprehension and retention of key HAZWOPER concepts, and how it supports you as trainers in presenting these materials more effectively.

DETAILED DESCRIPTION:
IMPRINT aims to enhance trainee performance and set operational expectations outside of the hot zone in hyper-realistic exercises that challenge physical, psychological, and cognitive capabilities through adaptive behavioral science enhanced VR modules and seamlessly integrate with HAZWOPER training.

The investigators anticipate trainees and classes assigned to the intervention will perform better than those who use standard paper and PowerPoint based activities. The investigators believe their comprehension of topics will be greater, and it is likely that they will have a greater ability to recall HAZWOPER guidelines in the field. The investigators also anticipate after class survey results will indicate a better HAZWOPER training experience and increased levels of satisfaction with the course.

Additionally, the investigators anticipate that trainers using the IMPRINT VR modules will find the tool more effective and engaging compared to standard PowerPoint and video-based training methods. The investigators expect that trainers will report greater ease in delivering complex HAZWOPER concepts and that the VR modules will enhance their ability to facilitate trainee comprehension and recall of HAZWOPER guidelines. We also anticipate that trainer feedback will reflect a more positive teaching experience and higher levels of satisfaction with the training process.

Long-term benefits of participation include improvement in retention of HAZWOPER guidelines when responding to Hazardous Material (HAZMAT) disasters. The investigators anticipate trainees and classes assigned to the intervention will perform better than those who use standard paper and PowerPoint based activities. The investigators believe their comprehension of topics will be greater, and it is likely that they will have a greater ability to recall HAZWOPER guidelines in the field. The investigators also anticipate after class survey results will indicate a better HAZWOPER training experience and increased levels of satisfaction with the course.

To successfully transfer skills and develop trainees' procedural cognitive maps VR training systems must enable full immersion into training exercises by integrating PPE, enabling 3D object haptic interaction and natural walking to support spatial skill development, and provide trainer support. Research has shown significant performance benefits from VR delivered targeted mission rehearsal. To realize these benefits before facing real emergencies, trainees must have the opportunity to hone their skills in a controlled setting that mimics real-life scenarios as closely as possible through fully immersive exercises. This immersive context driven approach is critical for skill transfer and well understood in parallel domains. Immersion is best achieved through a combination of sensations, including haptic (tactile touch, force feedback, temperature, etc.), audio, and visual (simulated detector reads of simulated radiation). Several recent empirical assessments of VR systems demonstrate superior skill transfer when haptic immersion is integrated in a domain appropriate way (e.g., heat exposure fire training, or stress inducing stimuli for disaster response).

It is not known whether this skill transfer occurs within the HAZMAT domain, or how to best operationalize these findings within training.

ELIGIBILITY:
The investigators will be targeting participants who participate in The New England Consortium (TNEC) training offerings. Given the training takes place in Massachusetts the investigators will use Massachusetts demographics to set our inclusion targets.

Inclusion Criteria:

* Students taking the 40-hr HAZWOPER course at The New England Consortium
* Trainers teaching the 40-hr HAZWOPER course at The New England Consortium

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: American Indian or Alaskan Native: .01% Asian: 9% Black or African American: 9.9% Hispanic or Latinx: 20.5% Native Hawaiian or other Islander: 0% Multiple Race, Non-Hispanic: 0% White: 56.7%
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
System Usability Scale | Immediately after the intervention
  SUS measures the usability of a system or interface. Higher scores on SUS indicate better usability. Typically, SUS scores are standardized to a scale of 0 to 100, where a score above 68 is considered above average usability, and scores above 80 indicate excellent usability
NASA TLX | Immediately after the intervention
  The NASA TLX is a scale from 0 - 100 and measures perceived workload across different domains such as mental demand, physical demand, temporal demand, performance, effort, and frustration. Higher NASA TLX scores indicate higher perceived workload, meaning that a lower score generally suggests a better outcome in terms of reduced workload. However, for this effort, we are specifically assessing whether the workload in VR aligns with the high workload typically experienced during an actual HAZWOPER incident

SECONDARY OUTCOMES:
User satisfaction with the VR modules | Post Study / after completing all interventions
  User satisfaction with the VR modules, evaluated through post-session surveys. This was accomplished as part of the debrief Q and A

CONTACTS AND LOCATIONS:
Locations (1):
- The New England Consortium, Lowell, Massachusetts, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-02): https://cdn.clinicaltrials.gov/large-docs/07/NCT06861907/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT06861907/ICF_001.pdf